CLINICAL TRIAL: NCT00932152
Title: A Phase II Randomized Trial of Fulvestrant and Anastrozole as Consolidation Therapy in Postmenopausal Women With Advanced Non-small Cell Lung Cancer Who Have Received First-line Platinum-based Chemotherapy With or Without Bevacizumab
Brief Title: Fulvestrant and Anastrozole as Consolidation Therapy in Postmenopausal Women With Advanced Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor enrollment/suspended to accrual; will close per AstraZeneca request
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Ahmad Tarhini, Associate Professor of Medicine and Translational Science, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPCI 08-131
Record Dates: First submitted 2009-07-01; First posted 2009-07-03 (Estimated); Results first posted 2016-08-31 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-09

CONDITIONS: Non-small Cell Lung Cancer; Postmenopausal Women
Keywords: advanced non-small cell lung cancer; postmenopausal; bevacizumab; fulvestrant; anastrozole
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Fulvestrant; Anastrozole; Bevacizumab; Anti-Bacterial Agents; Analgesics; Antiemetics; Thoracentesis; Pleurodesis; Blood Transfusion; Nutritional Support

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm B, Group 1 (Active Comparator): Best supportive care only: antibiotics, analgesics, antiemetics, thoracentesis, pleurodesis, blood transfusions, and/or nutritional support PRN
  Interventions: Drug: Best supportive care
- Arm B, Group 2 (Active Comparator): Best supportive care and Bevacizumab 15mg/kg every 21 days
  Interventions: Drug: Bevacizumab (Avastin); Drug: Best supportive care
- Arm A, Group 1 (Experimental): Fulvestrant and anastrozole only
  Interventions: Drug: fulvestrant (Faslodex); Drug: anastrozole (Arimidex)
- Arm A, Group 2 (Experimental): Fulvestrant, anastrozole and Bevacizumab
  Interventions: Drug: fulvestrant (Faslodex); Drug: anastrozole (Arimidex); Drug: Bevacizumab (Avastin)

INTERVENTIONS:
Drug: fulvestrant (Faslodex) — Fulvestrant (Faslodex) IM 250 mg monthly after a loading dose of 500 mg on day 1 and 250 mg on day 15 of cycle 1.
  Arms: Arm A, Group 1; Arm A, Group 2
Drug: anastrozole (Arimidex) — Anastrozole (Arimidex) 1 mg orally QD
  Arms: Arm A, Group 1; Arm A, Group 2
Drug: Bevacizumab (Avastin) — Bevacizumab (Avastin) 15 mg/kg IV, every 21 days
  Arms: Arm A, Group 2; Arm B, Group 2
Drug: Best supportive care — Subjects will not receive any chemotherapy for NSCLC nor will they received anti-cancer surgery, immunotherapy, radiotherapy or hormonal therapy. Among the therapies they may take are therapies considered acceptable include, but are not limited to, antibiotics, analgesics, antiemetics, thoracentesis, pleurodesis, blood transfusions, and/or nutritional support (enteral or parenteral
  Other Names: Antibiotics, analgesics, antiemetics, thoracentesis, pleurodesis, blood transfusions, and/or nutritional support
  Arms: Arm B, Group 1; Arm B, Group 2

SUMMARY:
This research study will test whether dual anti-estrogen therapy (anastrozole and fulvestrant) slows the time to when the cancer progresses.

DETAILED DESCRIPTION:
Women invited to participate in this study must be post-menopausal and be 18 years of age or older. The study is being performed on a total of 100 individuals. Of this group, 75 will be in the Treatment Groups using Fulvestrant/Anastrozole with our without bevacizumab and 25 will be in the "Best Supportive Care" groups receiving no treatment or just bevacizumab at the University of Pittsburgh Medical Center.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of non-small cell lung cancer (NSCLC) (no component of small cell).
* Patients must have stage IIIB (with malignant pleural effusion), stage IV NSCLC (as staged by the AJCC Cancer Staging Manual. 6th ed, appendix 1) or stage IV NSCLC as staged by the new AJCC staging system
* Patients with recurrent NSCLC should have recurred 12 months or more after completion of prior chemotherapy given in the context of curative therapy (chemoradiotherapy or adjuvant therapy) are eligible
* Patients should have been treated with 4 cycles of induction chemotherapy utilizing the following regimens: carboplatin/paclitaxel, carboplatin/gemcitabine, carboplatin/paclitaxel + bevacizumab, carboplatin/gemcitabine + bevacizumab, or carboplatin/pemetrexed +/- bevacizumab, (see Section 3.2 for acceptable doses and schedules) and should have CR, PR, or SD as best response.
* Patients should not have progressed on prior chemotherapy for metastatic or recurrent NSCLC.
* Must be postmenopausal female, as defined by the following criteria:

  * Prior bilateral oophorectomy or
  * Age greater than 60 years old
  * Age less than 60 years old and amenorrheic for 12 or more months in the absence of chemotherapy or ovarian suppression with FSH and estradiol in the postmenopausal range.
* Registration/randomization should be within 6 weeks of beginning of last cycle of chemotherapy
* Documented evidence of a tumor response of CR, PR, or SD. Tumor assessment must occur between Cycle 4 (Day 1) of induction therapy and the date of randomization. Tumor assessment will be per RECIST (Appendix 3) by the treating physician. This response does not have to be confirmed in order for the patient to be randomized; however, unconfirmed responses will be stratified in the stable disease strata. Positron emission tomography (PET) scans and ultrasound may not be used for lesion measurements for response determination
* ECOG performance status 0, 1 or 2.
* At least 18 years of age.
* Adequate organ function, including the following:

Adequate bone marrow reserve: absolute neutrophil (segmented and bands) count (ANC) greater than or equal to 1.0 x10^9/L, platelets greater than or equal to 75 x10^9/L, and hemoglobin greater than or equal to 9 g/dL.

Hepatic: bilirubin less than or equal to 1.5 times the upper limit of normal (ULN), alkaline phosphatase (ALP), aspartate transaminase (AST), and alanine transaminase (ALT) less than or equal to 2.0 Renal: calculated creatinine clearance (CrCl) ≥45 mL/min based on the standard Cockcroft and Gault formula (Cockcroft and Gault 1976).

* Prior radiotherapy must be completed at least 3 weeks before study enrollment. Patients must have recovered from the acute toxic effects of the treatment prior to study enrollment.
* Signed informed consent document on file.
* Patient compliance and geographic proximity that allow adequate follow up.
* Patient must receive on-study therapy no earlier than 21 days and no later than 42 days from their last cycle (Day 1) of induction therapy.
* Patients must have archival tissue samples. Tumor tissue will be submitted for assessment of ERa, ERb, PR, VEGF and aromatase expression. The patient must also agree to mandatory correlative blood samples at baseline, 5 weeks, 9 weeks, 13 weeks and at the time of progression.
* Cisplatin may be used instead of carboplatin as part of the initial induction chemotherapy regimen, at the discretion of the treating physician investigator. The dose and schedule of cisplatin will be according to the standard of care for patients with stage IIIB with malignant pleural effusion or stage IV NSCLC as staged by the AJCC Cancer Staging Manual, 6th ed, appendix 1, that is equivalent to stage IV NSCLC as staged by the new 7th ed AJCC staging system.

Exclusion Criteria:

* Male gender
* With the exception of those chemotherapies listed as Inclusion criterion (4) No other concomitant biological therapy (e.g. cetuximab) is allowed.
* Have received experimental treatment within the last 30 days at the time of study entry.
* Inability to comply with protocol or study procedures.
* A serious concomitant systemic disorder that, in the opinion of the investigator, would compromise the patient's ability to complete the study.
* Concurrent administration of any other antitumor therapy (except arm B, who are allowed to continue with bevacizumab).
* Pregnant or breast feeding.
* Have a prior malignancy other than NSCLC, carcinoma in situ of the cervix, or nonmelanoma skin cancer, unless that prior malignancy was diagnosed and definitively treated at least 5 years previously with no subsequent evidence of recurrence.
* Patients with two or more deep vein thromboses, or an active deep vein thrombosis.
* Patients taking hormone replacement therapy or other hormonal therapies
* The International Normalized Ratio (INR) must be < 1.6 within 28 days prior to registration.
* Patients with bleeding diathesis (i.e., disseminated intravascular coagulation [DIC], clotting factor deficiency) or a history of recent history of hemoptysis (1/2 tsp of red blood). Patients on stable long term anticoagulation prior to starting this trial are allowed.
* History of hypersensitivity to active or inactive excipients of fulvestrant (ie castor oil or Mannitol).
* Treatment of NSCLC with squamous cell histology with bevacizumab.
* No progressive Brain or CNS metastases
* No other concurrent anticancer therapy is allowed other than Bevacizumab

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2010-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Tarhini, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participants were randomized to the "Best supportive care only" and "Best supportive care with Bevacizumab" Arms due to low recruitment.
Period: Overall Study
Arm/Group | Fulvestrant and Anastrozole Only | Fulvestrant, Anastrozole and Bevacizumab
Started | 1 | 2
Completed | 0 | 0
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fulvestrant and Anastrozole Only | Fulvestrant, Anastrozole and Bevacizumab | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Continuous [Mean (Full Range); unit: years] | 67 [67 to 67] | 67.5 [58 to 77] | 67 [58 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate the Progression-free Survival.
Time Frame: 1.5 years
Population: Analysis was not completed because the trial was stopped prematurely due to slow accrual.
Arm/Group | All Participants (Overall Study)
Number analyzed (Participants) | 0

2. Secondary Outcome: To Evaluate the Time to Overall Survival, Time to Progression, and Toxicities
Time Frame: 1.5 years
Population: No data displayed because Outcome Measure has zero total participants analyzed.
Arm/Group | Fulvestrant and Anastrozole Only | Fulvestrant, Anastrozole and Bevacizumab
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: To Evaluate the Levels of 17b-estradiol, VEGF, E-selectin, Thrombospondin-1 and IGF-1, and Other Biomarkers in the Plasma.
Time Frame: 1.5 years
Population: No data displayed because Outcome Measure has zero total participants analyzed.
Arm/Group | Fulvestrant and Anastrozole Only | Fulvestrant, Anastrozole and Bevacizumab
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: To Evaluate Biomarkers (ERa, ERb, PR, VEGF and Aromatase Expression) in Baseline, Archival Tumor Tissue and Correlate Their Expression With Progression-free Survival, Time to Progression, and Overall Survival.
Time Frame: 1.5 years
Population: No data displayed because Outcome Measure has zero total participants analyzed.
Arm/Group | Fulvestrant and Anastrozole Only | Fulvestrant, Anastrozole and Bevacizumab
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Adverse events were not collected/monitored "per Arm/Group"
Arm/Group | All Participants (Overall Study)
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (Overall Study) (N=3)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Obstruction, GI, Small bowel NOS (Gastrointestinal disorders) | 1
Neurology - Other (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (Overall Study) (N=3)
Leukocytes (total WBC) (Investigations) | 1
Lymphopenia (Investigations) | 1
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 1
Hypertension (Vascular disorders) | 2
Fatigue (asthenia, lethargy, malaise) (General disorders) | 2
Rigors/chills (General disorders) | 1
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 1
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1
Hot flashes/flushes (Vascular disorders) | 2
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Mucositis/stomatitis (functional/symptomatic), Oral cavity (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils, Conjunctiva (Infections and infestations) | 1
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 1
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 1
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 1
Bilirubin (hyperbilirubinemia) (Investigations) | 1
Glomerular filtration rate (Renal and urinary disorders) | 1
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 2
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 1
Mood alteration, Depression (Psychiatric disorders) | 1
Neurology - Other (Nervous system disorders) | 1
Neuropathy: sensory (Nervous system disorders) | 1
Watery eye (epiphora, tearing) (Eye disorders) | 1
Pain, Abdomen NOS (Gastrointestinal disorders) | 1
Pain, Back (Musculoskeletal and connective tissue disorders) | 1
Pain, Extremity-limb (Musculoskeletal and connective tissue disorders) | 1
Pain, Head/headache (Nervous system disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1
Vaginal dryness (Reproductive system and breast disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes